CLINICAL TRIAL: NCT03336008
Title: Hong Kong Spinocerebellar Ataxias Registry
Acronym: HK_SCA_Reg
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Anne YY CHAN, Associate Consultant, Chinese University of Hong Kong
Other Study IDs: HK_SCA_Registry
Record Dates: First submitted 2017-09-29; First posted 2017-11-08 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Spinocerebellar Ataxia
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — No intervention but clinical assessement for all recruited subjects

SUMMARY:
Spinocerebellar ataxias (SCA) 1, 2, 3 and 6 are the most common, autosomal dominantly inherited cerebellar degenerations. And in the Chinese population, the most common SCA is SCA3 and the frequency of SCA 3 among SCA patients is 72.5%, followed by SCA 2 that the frequency is 12% among SCA patients. For SCA 1, the frequency among SCA patients is 7%. Even SCAs are rare diseases, a significant amount of Chinese in Hong Kong still suffer from this disorders. SCA Association in Hong Kong has 88 members who are suffering from spinocerebellar degeneration, many of them have a genetic confirmation. As there are few treatments for SCAs; therefore, understanding SCAs clinical manifestation and disease mechanisms are the first step towards development of effective treatment. The objective of this study is to develop the first SCA registry in Hong Kong with bio-repository bank for clinical and genetic information as well as serum and fibroblasts.

DETAILED DESCRIPTION:
All the members from Hong Kong SCA association will be invited and discuss the study with them. After obtaining the informed consent, their genotypes will be determined and collect clinical information. Some of the participant will have clear genotyping via Department of Health. Participants with a genetic confirmation of SCA1, 2, 3, 6, 7, 8 and 12 genes will be included in the study. The relatives of genetically confirmed participants, who also had ataxic symptoms, might be included in the study without further determination of the genotypes.

Detailed clinical history including age of onset, clinical symptoms will be collected. A detailed neurological examination with an emphasis of eye movements (such as pursuit, saccadic, and convergence eye movements). We will also perform SARA scale, a validated ataxia scale. Timed 25 foot-walk test will be performed.

Two-year annual follow-up will be arranged for recruited subject for neurological physical examination, SARA scale, in order to continue assessment for any progress change in disease stage.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above
2. Presence of symptoms and signs of ataxia
3. Definite molecular diagnosis of SCA1, 2, 3, 6, 7, 8 or 12 either in the participant or another affected family member
4. Willingness to participate in the study and ability to give informed consent

Exclusion Criteria:

1. Known recessive. X-linked, and mitochondrial ataxias

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SCA association members or SCA subjects who follow-up in our clinic or refer from other clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-12-07 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Scale for the assessment and rating of ataxia (SARA) score | change from baseline to 2-year follow up
  Scale for the assessment and rating of ataxia (total score 0-40)

SECONDARY OUTCOMES:
EQ5D Health questionnaire | change from baseline to 2-year follow up
  EQ-5D is a standardized instrument for measuring generic health status. The health status measured with EQ-5D is used for estimating preference weight for that health status (1-3 in each health status , 0-100 in general today's health status)
Patient Health Questionnaire-9 (PHQ-9) | change from baseline to 2-year follow up
  Depression scale (0-4 in each items)

CONTACTS AND LOCATIONS:
Overall Officials: Anne YY CHAN, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No